CLINICAL TRIAL: NCT05055856
Title: Asymptomatic Bacteriuria, Hyponatremia and Geri-atric Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: asymptomatische bacteriuria
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Asymptomatic Bacteriuria; Frailty; Geriatric Syndrome; SIADH
MeSH Terms: conditions — Frailty; Inappropriate ADH Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: academic, prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frailty or more (Active Comparator): patients with the geriatric syndrome who will be recruited at the geriatric out patient clinic
  Interventions: Diagnostic Test: urine sample; Diagnostic Test: Blood and urine sample
- healthy (Placebo Comparator): healthy aged people defined as in the modified SENIEUR protocol who will be recruited by an extern call thanks UZ Brussel website of thanks to staff's knowledge
  Interventions: Diagnostic Test: urine sample; Diagnostic Test: Blood and urine sample

INTERVENTIONS:
Diagnostic Test: urine sample — Each participant will give a urine sample for diagnose of asymptomatic bacteriuria
Diagnostic Test: Blood and urine sample — Each participant will give a urine and blood sample for diagnose of SIADH

SUMMARY:
The population is aging. Aged people are more prown to develop frailty. The causes of frailty are multifactorial and are being investigated in research settings. Cardiovascular diseases, inflammaging and changes in microbiota have been associated with frailty and geriatric syndrome. The prevalence of asymptomatic bacteriuria and SIADH-related hyponatremia is also important in aging and associated with inflammaging. The aim of this study is to examine, if asymptomatic bacteriuria and SIADH-related hyponatremia could be markers for frailty and geriatric syndrome.

DETAILED DESCRIPTION:
The demographic evolution represents a challenge for the general public health. The global population, especially in the developed countries, is aging. Aging is associated with a decrease of physio-logical functions leading to frailty. Frailty is an important concept in geriatric medicine: it is a biological syndrome of decreased reserve and resistance to stressors resulting from cumulative decline across multiple physiological systems (like osteopenia, sarcopenia, dysregulation of hypothalamic axis …). Factors that lead to frailty influence each other and can be self-perpetuating. Frailty is a geriatric syndrome but there are a lot of other geriatric syndrome such as falls, undernutrition,… When young people are sick, they present mostly more than one symptom who can be referred to one disease or one cause. In contrast, geriatric patients will present one symptom, such as confusion, fall, undernutrition,… which can be referred to multifactorial causes or diseases. This is the concept of geriatric syndrome.

Frailty or geriatric syndrome has been related to inflammaging. Inflammaging, characterized by an increase of circulating cytokines such as interleukin (IL)-6 and acute phase proteins, is a feature of immunosenescence. This process of immunosenescence is suggested to participate in the pathogene-ses of frailty and geriatric syndromes. The possible origins of inflammaging are multifactorial and controversies still exist: cardiovascular (CV) diseases, depression and chronic cytomegalovirus (CMV) infections are associated with this pro-inflammatory state. These comorbidities are highly prevalent in geriatric patients and could therefore contribute to the association between low-grade inflammation, frailty and geriatric syndromes.

The intestinal barrier and microbiota are associated with frailty and inflammaging. Multiple potential pathways exist through which the gut microbiota can provoke inflammaging (through TLR, stimulation of immune cells, translocation, endotoxines et cetera). In the same way of thinking, asymptomatic bacteriuria could also be responsible of inflammaging and frailty. The prevalence of asymptomatic bacteriuria is increased with aging and in patient with diabetes. It has also been shown to be associated with chronic inflammation (sTNFR and TNFα), increased WBCC and neutrophils. To our knowledge, it is unknown if asymptomatic bacteriuria is associated with frailty.

Hyponatremia is highly prevalent in hospitalized patients. SIADH-related hyponatremia represents 1/3 of the causes of hyponatremia. The incidence of SIADH related hyponatremia is believed to be higher in older people. It is associated with an increased risk of falls, confusion and mortality. The physiological balance between water and salt changes with aging. SIADH is classified as an euvo-lemic status; however, it is caused by an excess of water. The inappropriate secretion of vasopressin( ADH=anti-diuretic hormone) increases the expression of the aquaporins in the renal tubules. These aquaporines increase the reabsorption of water resulting in an altered ratio of reabsorption of water and Salt, leading to hyponatremia. SIADH-related hyponatremia is also associated with inflammation. IL-6 and IL-1β are able to stimulate the pituitary-hypothalamic axis to secrete vasopressin. SIADH related hyponatremia could be also a sign of inflammaging and related with frailty.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years old
* Informed consent
* Presence of the geriatric syndrome (dementia, depression, frailty, dependence, fall, undernu-trition, incontinence…) or not in function of the group

Exclusion Criteria:

* Symptoms of urinary tract infection
* Confusion
* CRP > 5 mg/L
* Previous urological history
* Intake of antibiotics
* Intake of diuretics
* Intake of SSRI

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
asymptomatic bacteriuria | At baseline
  If the presence of an asymptomatic bacteriuria is associated with frailty or the geriatric syn-drome
SIADH | At baseline
  If the presence of SIADH-related hyponatremia is associated with frailty or geriatric syn-drome
SIADH and inflammaging | At baseline
  If the presence of SIADH-related hyponatremia is associated with a low grade chronic in-flammation as demonstrated by a raised c-reactive protein (CRP).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Compte, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fulop T, Witkowski JM, Olivieri F, Larbi A. The integration of inflammaging in age-related diseases. Semin Immunol. 2018 Dec;40:17-35. doi: 10.1016/j.smim.2018.09.003. Epub 2018 Oct 2. PMID 30287177
- [Background] Prio TK, Bruunsgaard H, Roge B, Pedersen BK. Asymptomatic bacteriuria in elderly humans is associated with increased levels of circulating TNF receptors and elevated numbers of neutrophils. Exp Gerontol. 2002 May;37(5):693-9. doi: 10.1016/s0531-5565(02)00002-5. PMID 11909686
- [Background] Swart RM, Hoorn EJ, Betjes MG, Zietse R. Hyponatremia and inflammation: the emerging role of interleukin-6 in osmoregulation. Nephron Physiol. 2011;118(2):45-51. doi: 10.1159/000322238. Epub 2010 Dec 22. PMID 21196778
- [Background] Bergsten G, Wullt B, Svanborg C. Escherichia coli, fimbriae, bacterial persistence and host response induction in the human urinary tract. Int J Med Microbiol. 2005 Oct;295(6-7):487-502. doi: 10.1016/j.ijmm.2005.07.008. PMID 16238023